CLINICAL TRIAL: NCT01790633
Title: Pilot Study Evaluating the Use of Simultaneous HBV, HCV, and HIV Rapid Tests As a Tool for Screening and Access to Care Among At-Risk Populations
Brief Title: Pilot Study Evaluating the Use of Simultaneous HBV, HCV, and HIV Rapid Tests
Acronym: OPTISCREEN-III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government); Gilead Sciences (Industry); Roche Pharma AG (Industry); Mairie de Paris (Unknown); BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IMEA 38B; 2012-A01681-42 (Other: ANSM)
Record Dates: First submitted 2013-02-07; First posted 2013-02-13 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-10

CONDITIONS: HIV; Hepatitis B; Hepatitis C; Carcinoma, Hepatocellular; AIDS
Keywords: rapid test; screening; ELISA; hepatitis B virus; hepatitis C virus; human immunodeficiency virus; access to care
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Carcinoma, Hepatocellular; Acquired Immunodeficiency Syndrome | interventions — Enzyme-Linked Immunosorbent Assay; Rapid Diagnostic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard testing with ELISA (Active Comparator): HBV, HCV, and HIV infection status determined by enzyme-linked immuno-assay (ELISA).
  Interventions: Other: ELISA
- Rapid testing (Experimental): HBV, HCV, and HIV infection status determined by a rapid test
  Interventions: Other: Rapid Test

INTERVENTIONS:
Other: ELISA — Enzyme-linked immuno-assay (ELISA) will be used to determine hepatitis B surface antigen (HBsAg), anti-HBsAg antibody (anti-HBs Ab), anti-HCV antibody, and anti-HIV antibody status. Results will be given after test results are available (8-10 days).
  Arms: Standard testing with ELISA
Other: Rapid Test — A rapid test will be performed to determine the subjects' hepatitis B surface antigen (HBsAg, using VIKIA®), anti-HCV antibody (HCV, using OraQuick®), and anti-HIV antibody (HIV, using VIKIA®) status. Results will be given the same day.
  Other Names: VIKIA®, Biomerieux, Marcy-l'Étoile, France; OraQuick® HCV Rapid Antibody Test, OraSure Technologies, Inc., Bethlehem, PA, USA
  Arms: Rapid testing

SUMMARY:
This is a pilot, monocentric, prospective, randomized control trial looking at the use of rapid tests as a part of normal care. The investigators will be testing for hepatitis B virus (HBV), hepatitis C virus (HCV), and human immunodeficiency virus (HIV). Testing will be proposed to all persons seeking care at the Centre d'Accueil, de Soins et d'Orientation from the organization Médecin du Monde (CASO, MDM).

Infection status of participants will be determined by either the standard test (ELISA) or rapid test. The choice between tests will be determined randomly.

The overall goal is to determine the general acceptability and feasibility of rapid tests and to see if they can help individuals increase their awareness of infection status when compared to longer, routine methods of testing. In addition, results from these tests will allow the medical doctor to guide participants to appropriate care. All positive tests will be confirmed at a specialized hospital (Hôptial Saint-Antoine, Paris, France) and health-specific information will be obtained four months after testing.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Seeking care at the CASO MDM health care center
* Accept to be followed at Saint-Antoine Hospital in the event of a positive test.

Exclusion Criteria:

* Currently under physician's care for viral hepatitis (HBV/HCV-specific) or HIV
* Already has been tested (must give any of the following as evidence):

  * results from HBV and HCV and HIV tests dating at least 3 months back
  * results from HCV and HIV tests dating at least 3 months back and HBV serology indicating that the participant is immunized against HBV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bottero, MD, Principal Investigator — Hôpital Saint-Antoine
Locations (1):
- Consultation d'Accueil, de Soins et d'Orientation (CASO) de Médecins du Monde (MDM), Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared under the following conditions: (1) interested parties must submit a request for data access to the principal investigator and (2) the request is approved by the Scientific Committee.

REFERENCES:
- [Background] Bottero J, Boyd A, Gozlan J, Lemoine M, Carrat F, Collignon A, Boo N, Dhotte P, Varsat B, Muller G, Cha O, Picard O, Nau J, Campa P, Silbermann B, Bary M, Girard PM, Lacombe K. Performance of rapid tests for detection of HBsAg and anti-HBsAb in a large cohort, France. J Hepatol. 2013 Mar;58(3):473-8. doi: 10.1016/j.jhep.2012.11.016. Epub 2012 Nov 23. PMID 23183527
- [Result] Bottero J, Boyd A, Gozlan J, Carrat F, Nau J, Pauti MD, Rougier H, Girard PM, Lacombe K. Simultaneous Human Immunodeficiency Virus-Hepatitis B-Hepatitis C Point-of-Care Tests Improve Outcomes in Linkage-to-Care: Results of a Randomized Control Trial in Persons Without Healthcare Coverage. Open Forum Infect Dis. 2015 Oct 26;2(4):ofv162. doi: 10.1093/ofid/ofv162. eCollection 2015 Dec. PMID 26668814

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers were recruited from an innercity clinic for persons without healthcare coverage ("Médecins du Monde", Paris, France). From February 25, 2013 to June 21, 2013, individuals seeking care at the center were asked to participate.
Pre-assignment Details: 554 participants were initially screened for eligibility. 150 did not meet inclusion criteria, 16 had a medical condition requiring immediate referral to a specialist, and 61 declined to participate. A total of 327 were randomized.
Period: Overall Study
Arm/Group | Standard Testing With ELISA | Rapid Testing
Started | 163 | 164
Completed | 115 | 159
Not Completed | 48 | 5
Not completed — Protocol Violation | 1 | 2
Not completed — Did not have serology performed | 47 | 0
Not completed — RT failure and no follow-up ELISA | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Testing With ELISA | Rapid Testing | Total
Number analyzed (Participants) | 162 | 162 | 324
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (12.2) | 37.0 (12.2) | 37.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 63 | 123
  Male | 102 | 99 | 201
HBV prevalence of birth country [Number; unit: participants]
  Low (<2.0%) | 2 | 1 | 3
  Intermediate (2.0%-8.0%) | 27 | 37 | 64
  High (>8.0%) | 133 | 124 | 257
No health insurance plan [Number; unit: participants] | 162 | 162 | 324

OUTCOME MEASURES:

1. Primary Outcome: Accessibility of Testing Results
Description: The number of individuals who obtained test results for HBV, HCV, and/or HIV divided by the total number of tested individuals.
Time Frame: Evaluated once, up to 4 months after testing
Measure: Number; unit: proportion of participants
Arm/Group | Standard Testing With ELISA | Rapid Testing
Number analyzed (Participants) | 162 | 162
proportion of participants | 0.642 | 0.981
Statistical Analysis 1: Comparison: Standard Testing With ELISA vs Rapid Testing; We approached our analysis as a pilot study with the aim of addressing feasibility. 70% of patients seen at the MDM clinic obtain a test result with standard serology. Assuming a 20% increase in infection awareness and type 1 error of 0.05, and power of at least 0.9, a minimum of 82 participants per group would be needed; Test type: Superiority or Other; p < 0.001, Chi-squared — P-value adjustments for multiple comparisons were not necessary. Significance was determined using P < 0.05

2. Secondary Outcome: Access to Care
Description: The number of individuals seeking specialized care with a complete evaluation of disease severity divided by the total number of seropositive individuals.
Time Frame: Evaluated once, up to 4 months after testing
Population: Analysis includes only participants with positive HIV, HBV, and/or HCV results.
Measure: Number; unit: proportion of participants
Arm/Group | Standard Testing With ELISA | Rapid Testing
Number analyzed (Participants) | 16 | 20
proportion of participants | 0.938 | 0.900
Statistical Analysis 1: Comparison: Standard Testing With ELISA vs Rapid Testing; Test type: Superiority or Other; p = 0.7, Chi-squared — P-value adjustments for multiple comparisons were not necessary. Significance was determined using P < 0.05

3. Other Pre Specified Outcome: Proportion Participating
Description: The number of individuals accepting to participate in the study divided by the total number of individuals proposed.
Time Frame: At testing
Measure: Number; unit: proportion of participants
Groups:
- Screened for Eligibility: Individuals who were screened for eligibility, prior to being considered for randomization.
Arm/Group | Screened for Eligibility
Number analyzed (Participants) | 554
proportion of participants | 0.890

4. Other Pre Specified Outcome: Proportion of Rapid Test Failures
Description: The number of rapid tests giving inconclusive results divided by the total number of rapid tests (only available in the rapid test arm).
Time Frame: At testing
Population: Only patients randomized to the rapid testing arm.
Measure: Number; unit: proportion of participants
Arm/Group | Standard Testing With ELISA | Rapid Testing
Number analyzed (Participants) | 0 | 162
proportion of participants |  | 0.074

ADVERSE EVENTS:
Arm/Group | Standard Testing With ELISA | Rapid Testing
Serious Adverse Events (participants affected / at risk) | 0/162 | 0/162
Other Adverse Events (participants affected / at risk) | 0/162 | 0/162

LIMITATIONS AND CAVEATS:
Single-center pilot study, possibly reducing generalizability; small number of participants and infected individuals may have decreased power to detect differences in linkage-to-care; not all rapid tests were approved for routine use in France.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No